CLINICAL TRIAL: NCT02093221
Title: A Multicenter, Randomized, Partial-Blinded, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a Human Plasma-Derived Alpha1-Proteinase Inhibitor in Subjects With New-Onset Type 1 Diabetes Mellitus
Brief Title: Study of Human Plasma-Derived Alpha1-Proteinase Inhibitor in Subjects With New-Onset Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Wk 52 primary endpoint results would be unaffected by follow-up data so trial was discontinued prior to wk 104. No safety data was collected after wk 52.
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTI1302
Record Dates: First submitted 2014-03-11; First posted 2014-03-20 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Alpha1-Proteinase Inhibitor; Beta Cell; Alpha1-Antitrypsin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin; Mp alpha1 receptor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Alpha1-PI 180 mg/kg/wk, 26 weeks (Experimental): 180 mg/kg weekly infusions of Alpha1-PI for 26 weeks.
  Interventions: Biological: 180 mg/kg Alpha1-PI
- 90 mg/kg/wk Alpha1-PI, 26 weeks (Experimental): 90 mg/kg weekly infusions of Alpha1-PI for 26 weeks.
  Interventions: Biological: 90 mg/kg Alpha1-PI
- Placebo, 26 weeks (Placebo Comparator): Weekly infusions of placebo for 26 weeks.
  Interventions: Biological: Placebo
- 180 mg/kg/wk Alpha1-PI, 13 weeks (Experimental): 180 mg/kg weekly infusions of Alpha1-PI for 13 weeks.
  Interventions: Biological: 180 mg/kg Alpha1-PI
- 90 mg/kg/wk Alpha1-PI, 13 weeks (Experimental): 90 mg/kg weekly infusions of Alpha1-PI for 13 weeks
  Interventions: Biological: 90 mg/kg Alpha1-PI
- Placebo, 13 weeks (Placebo Comparator): Weekly infusions of placebo for 13 weeks.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 180 mg/kg Alpha1-PI
  Other Names: Alpha1-antitrypsin; Prolastin-C; Alpha1-Proteinase Inhibitor (human), Modified Process; Alpha-1 MP
  Arms: 180 mg/kg/wk Alpha1-PI, 13 weeks; Alpha1-PI 180 mg/kg/wk, 26 weeks
Biological: 90 mg/kg Alpha1-PI
  Other Names: Alpha1-antitrypsin; Prolastin-C; Alpha1-Proteinase Inhibitor (human), Modified Process; Alpha-1 MP
  Arms: 90 mg/kg/wk Alpha1-PI, 13 weeks; 90 mg/kg/wk Alpha1-PI, 26 weeks
Biological: Placebo
  Arms: Placebo, 13 weeks; Placebo, 26 weeks

SUMMARY:
This is a multicenter, randomized, partial-blinded, five-arm, placebo-controlled study of human plasma-derived alpha1-proteinase inhibitor (alpha1-PI) in children (ages 6-11 years old) and teens/adults (ages 12-35 years old) with new onset Type 1 Diabetes Mellitus (T1DM). Currently enrolling ages 12-35 only. Once 25 patients are randomized and data is reviewed enrollment will be opened to the child cohort. The purpose of this study is to evaluate the safety and efficacy of four dosing regimens of human plasma-derived alpha1-PI in T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1DM according to the ADA criteria.
* Current use of injected insulin therapy and one positive result on testing for any of the following antibodies (If not currently on insulin therapy, must have positive result for at least two of the below antibodies):

  * Anti-islet-cell antibodies (islet cell antigen 512, insulinoma associated protein 2),
  * Anti-glutamic acid decarboxylase antibodies, or
  * Anti-insulin antibodies (unless received insulin therapy for > 7 days).
* Body Mass Index (BMI) ≤ 28 kg/m2 for adults (≥ 20 years of age) OR ≤ 90th percentile in accordance with the Centers for Disease Control BMI assessment for children and teens (2 through 19 years old).

Exclusion Criteria:

* History of or current diabetic retinopathy, neuropathy, or nephropathy.
* Known thrombophilia or history of thrombosis.
* Malignant disease (including malignant melanoma; however, other forms of skin cancer are allowed) within five years of randomization.
* Active Hepatitis A virus, Hepatitis B virus, Hepatitis C virus, or Human Immunodeficiency Virus infection.
* History of anaphylaxis or severe systemic response to any plasma-derived alpha1-PI preparation or other blood product(s).
* Known selective or severe Immunoglobulin A deficiency.
* Elevated liver enzymes (aspartate transaminase, alanine aminotransferase, and alkaline phosphatase) equal to or greater than 2.5 times the upper limit of normal.
* Therapy with exenatide or any other agents that stimulate pancreatic β cell regeneration or insulin secretion, or any antidiabetic agents (oral or parenteral) other than insulin within one month prior to screening.
* Use of omega-3 fatty acid supplements, including fish oil, within seven days prior to screening.
* Current or planned therapy with inhaled insulin, if it becomes available.
* Chronic use of systemic steroids, with the exception of inhaled steroids, above a stable dose equivalent to 5 mg/day prednisone (e.g., 10 mg every 2 days) within 4 weeks prior to randomization. It is recommended to maintain the same dose throughout the study. (Note: Subjects with autoimmune conditions (i.e., asthma) necessitating treatment with systemic short-term corticosteroids and administered a rapid taper are eligible per protocol with the caveat that the tapering is complete or decreased to the minimum requirement (i.e., 5 mg/day) at least 1 week prior to the Baseline visit (when randomization occurs) to ensure the subject is stable. For longer term steroid usage, please consult the Grifols Medical Monitor before considering the subject for study participation.)
* Treatment with immunosuppressants or cytostatic agents within 6 months of randomization.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - University of Arizona, Tucson, Arizona
  - Clinica Medica San Miguel, Los Angeles, California
  - Diabetes Associates Medical Group, Orange, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Metabolic Institute of America, Tarzana, California
  - Ronald H Chochinov MD, Ventura, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Solutions Through Advanced Research Inc., Jacksonville, Florida
  - CCM Clinical Research, Miami, Florida
  - Advanced Pharma CR LLC, Miami, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Cook County Hospital, Chicago, Illinois
  - Methodist Research Institute, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Barry J. Reiner MD, LLC., Baltimore, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - University of New Mexico, Health Sciences Center, Albuquerque, New Mexico
  - Women and Children's Hospital, Buffalo, New York
  - WakeMed Children's Hospital, Raleigh, North Carolina
  - Endocrinology Associates Inc, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Pediatric Endocrinology, Genetics & Metabolism, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rapid City Regional Hospital/Health Clinical Research, Rapid City, South Dakota
  - Research Institute of Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Northeast Clinical Research of San Antonio LLC, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Consano Clinical Research, San Antonio, Texas

REFERENCES:
- [Derived] Lagarde WH, Courtney KL, Reiner B, Steinmann K, Tsalikian E, Willi SM. Human plasma-derived alpha1 -proteinase inhibitor in patients with new-onset type 1 diabetes mellitus: A randomized, placebo-controlled proof-of-concept study. Pediatr Diabetes. 2021 Mar;22(2):192-201. doi: 10.1111/pedi.13162. Epub 2020 Dec 13. PMID 33244872

RESULTS

PARTICIPANT FLOW:
Groups:
- Alpha1-PI 180 mg/kg/wk, 26 Weeks: 180 mg/kg weekly infusions of Alpha1-PI for 26 weeks.
  180 mg/kg Alpha1-PI
- 180 mg/kg/wk Alpha1-PI, 13 Weeks: 180 mg/kg weekly infusions of Alpha1-PI for 13 weeks.
  180 mg/kg Alpha1-PI
- 90 mg/kg/wk Alpha1-PI, 26 Weeks: 90 mg/kg weekly infusions of Alpha1-PI for 26 weeks.
  90 mg/kg Alpha1-PI
- 90 mg/kg/wk Alpha1-PI, 13 Weeks: 90 mg/kg weekly infusions of Alpha1-PI for 13 weeks
  90 mg/kg Alpha1-PI
- Placebo: Weekly infusions of placebo for 13 or 26 weeks.
  Placebo
Period: Overall Study
Arm/Group | Alpha1-PI 180 mg/kg/wk, 26 Weeks | 180 mg/kg/wk Alpha1-PI, 13 Weeks | 90 mg/kg/wk Alpha1-PI, 26 Weeks | 90 mg/kg/wk Alpha1-PI, 13 Weeks | Placebo
Started | 15 | 16 | 15 | 15 | 15
Completed | 5 | 8 | 6 | 7 | 7
Not Completed | 10 | 8 | 9 | 8 | 8
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 4 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Study termination | 6 | 5 | 4 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpha1-PI 180 mg/kg/wk, 26 Weeks | 180 mg/kg/wk Alpha1-PI, 13 Weeks | 90 mg/kg/wk Alpha1-PI, 26 Weeks | 90 mg/kg/wk Alpha1-PI, 13 Weeks | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 15 | 15 | 15 | 76
Age, Customized [Count of Participants; unit: Participants]
  6 - 11 years | 2 | 3 | 3 | 3 | 2 | 13
  12 - 17 years | 7 | 7 | 7 | 7 | 6 | 34
  18 - 35 years | 6 | 6 | 5 | 5 | 7 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 9 | 4 | 4 | 31
  Male | 9 | 8 | 6 | 11 | 11 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 3 | 2 | 0 | 9
  Not Hispanic or Latino | 12 | 15 | 12 | 13 | 15 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 2 | 0 | 3
  White | 14 | 14 | 15 | 13 | 15 | 71
  More than one race | 1 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mixed Meal Tolerance Test (MMTMT) Stimulated C-peptide 2 Hour Area Under the Concentration-time Curve (AUC)
Description: C-peptide concentration during MMTT with high protein energy drink. "Dose" for time frame refers to intake of high protein energy drink.
Time Frame: Baseline, Week 52 (pre-high protein drink and 15, 30, 60, 90, 120 minutes post-drink)
Population: Twelve subjects prematurely discontinued from the study prior to Week 52.
Measure: Mean (Standard Deviation); unit: min*nmol/L
Arm/Group | Alpha1-PI 180 mg/kg/wk, 26 Weeks | 180 mg/kg/wk Alpha1-PI, 13 Weeks | 90 mg/kg/wk Alpha1-PI, 26 Weeks | 90 mg/kg/wk Alpha1-PI, 13 Weeks | Placebo
Number analyzed (Participants) | 13 | 14 | 11 | 12 | 14
min*nmol/L | -32.357 (27.7184) | -25.171 (28.9450) | -21.682 (24.5787) | -34.393 (25.6837) | -16.909 (19.1278)

2. Secondary Outcome: Change From Baseline for MMTT Stimulated C-peptide 2h AUC
Time Frame: Baseline, Weeks 14, 27, 39, 69, 87, and 104 (pre-high protein drink and 15, 30, 60, 90, 120 minutes post-drink)
Population: Forty-three subjects prematurely discontinued (prior to Week 104); 28 subjects were considered a premature discontinuation due to sponsor termination of the study.
Measure: Mean (Standard Deviation); unit: min*nmol/L
Arm/Group | Alpha1-PI 180 mg/kg/wk, 26 Weeks | 180 mg/kg/wk Alpha1-PI, 13 Weeks | 90 mg/kg/wk Alpha1-PI, 26 Weeks | 90 mg/kg/wk Alpha1-PI, 13 Weeks | Placebo
Number analyzed (Participants) | 15 | 16 | 15 | 15 | 15
min*nmol/L
  Week 14: number analyzed (Participants) | 12 | 13 | 14 | 14 | 14
  Week 14 | -19.396 (23.7789) | -0.444 (18.8595) | 4.427 (33.2220) | -12.725 (20.2051) | 3.317 (21.1784)
  Week 27: number analyzed (Participants) | 12 | 12 | 13 | 13 | 13
  Week 27 | -30.709 (21.2821) | -17.826 (21.0462) | 6.537 (56.1336) | -23.082 (22.3027) | -1.411 (26.8550)
  Week 39: number analyzed (Participants) | 10 | 10 | 10 | 12 | 12
  Week 39 | -28.500 (37.6682) | -17.664 (26.1729) | -23.342 (21.6945) | -36.580 (20.7765) | -10.808 (20.0078)
  Week 69: number analyzed (Participants) | 10 | 11 | 9 | 13 | 14
  Week 69 | -45.316 (27.1563) | -42.014 (15.7239) | -27.023 (28.6920) | -39.735 (23.3488) | -16.744 (21.8947)
  Week 87: number analyzed (Participants) | 7 | 11 | 7 | 10 | 9
  Week 87 | -42.487 (31.9418) | -43.012 (23.2403) | -34.590 (21.6148) | -47.496 (23.7717) | -32.561 (20.0826)
  Week 104: number analyzed (Participants) | 5 | 8 | 5 | 6 | 7
  Week 104 | -29.687 (25.5941) | -44.314 (28.0612) | -32.980 (18.2765) | -39.908 (26.4652) | -26.586 (20.6803)

3. Secondary Outcome: Change From Baseline for HbA1c Levels
Time Frame: Baseline, Weeks 14, 27, 39, 52, 69, 87, and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Alpha1-PI 180 mg/kg/wk, 26 Weeks | 180 mg/kg/wk Alpha1-PI, 13 Weeks | 90 mg/kg/wk Alpha1-PI, 26 Weeks | 90 mg/kg/wk Alpha1-PI, 13 Weeks | Placebo
Number analyzed (Participants) | 15 | 16 | 15 | 15 | 15
percentage of change from baseline
  Week 14: number analyzed (Participants) | 13 | 13 | 14 | 13 | 14
  Week 14 | -0.68 (2.108) | -1.75 (2.543) | -1.16 (1.683) | -1.45 (1.812) | -2.64 (2.452)
  Week 27: number analyzed (Participants) | 13 | 12 | 14 | 14 | 13
  Week 27 | -0.67 (1.953) | -1.38 (2.799) | -0.74 (2.263) | -0.89 (2.740) | -2.52 (2.439)
  Week 39: number analyzed (Participants) | 11 | 12 | 11 | 13 | 13
  Week 39 | -0.58 (2.098) | -0.78 (3.043) | -0.40 (1.495) | -0.55 (2.798) | -1.52 (2.473)
  Week 52: number analyzed (Participants) | 13 | 14 | 11 | 14 | 14
  Week 52 | -0.47 (1.383) | -0.55 (3.437) | -0.25 (1.399) | -0.51 (2.504) | -1.52 (2.805)
  Week 69: number analyzed (Participants) | 11 | 13 | 10 | 13 | 13
  Week 69 | -0.01 (1.630) | -0.18 (2.529) | 0.09 (1.197) | -0.33 (2.532) | -1.37 (3.004)
  Week 87: number analyzed (Participants) | 7 | 11 | 8 | 11 | 9
  Week 87 | -0.54 (1.310) | -0.38 (3.035) | 0.30 (2.147) | -0.26 (2.608) | -0.89 (3.011)
  Week 104: number analyzed (Participants) | 5 | 8 | 6 | 7 | 7
  Week 104 | -0.76 (1.419) | -0.69 (2.490) | 0.28 (1.987) | -0.10 (2.890) | -1.36 (2.155)

4. Secondary Outcome: Number of Subjects With Overall Severe Hypoglycemic Episodes
Description: Severe hypoglycemia defined according the ADA Workgroup on Hypoglycemia definition, as follows: An event requiring assistance of another person to actively administer carbohydrate, glucagons, or other resuscitative actions.
Time Frame: 104 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha1-PI 180 mg/kg/wk, 26 Weeks | 180 mg/kg/wk Alpha1-PI, 13 Weeks | 90 mg/kg/wk Alpha1-PI, 26 Weeks | 90 mg/kg/wk Alpha1-PI, 13 Weeks | Placebo
Number analyzed (Participants) | 15 | 16 | 15 | 15 | 15
Participants
  1 episode | 1 | 2 | 0 | 0 | 1
  2 episodes | 0 | 0 | 0 | 0 | 0
  3 episodes | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Change From Baseline for Mean Daily Insulin Dose Requirements
Time Frame: Baseline, Weeks 2, 4, 14, 27, 39, 52, 69, 87, and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | Alpha1-PI 180 mg/kg/wk, 26 Weeks | 180 mg/kg/wk Alpha1-PI, 13 Weeks | 90 mg/kg/wk Alpha1-PI, 26 Weeks | 90 mg/kg/wk Alpha1-PI, 13 Weeks | Placebo
Number analyzed (Participants) | 15 | 16 | 15 | 15 | 15
U/kg/day
  Week 2: number analyzed (Participants) | 8 | 9 | 7 | 7 | 9
  Week 2 | -0.146 (0.2044) | -0.141 (0.2143) | -0.205 (0.2194) | -0.274 (0.1416) | -0.158 (0.2828)
  Week 4: number analyzed (Participants) | 8 | 8 | 9 | 7 | 8
  Week 4 | -0.147 (0.1405) | -0.264 (0.1456) | -0.201 (0.2058) | -0.220 (0.1744) | -0.150 (0.2788)
  Week 14: number analyzed (Participants) | 9 | 7 | 7 | 7 | 8
  Week 14 | -0.239 (0.2301) | -0.305 (0.1406) | -0.092 (0.1442) | -0.239 (0.1430) | -0.118 (0.1114)
  Week 27: number analyzed (Participants) | 5 | 6 | 8 | 4 | 5
  Week 27 | -0.040 (0.2313) | -0.033 (0.4310) | -0.090 (0.2117) | -0.138 (0.2321) | -0.135 (0.0607)
  Week 39: number analyzed (Participants) | 3 | 5 | 8 | 5 | 4
  Week 39 | -0.040 (0.3222) | 0.146 (0.7900) | -0.089 (0.2099) | -0.158 (0.2552) | -0.150 (0.1100)
  Week 52: number analyzed (Participants) | 5 | 6 | 8 | 5 | 4
  Week 52 | 0.226 (0.5861) | -0.037 (0.8720) | -0.055 (0.2180) | 0.214 (0.5898) | -0.320 (0.2906)
  Week 69: number analyzed (Participants) | 3 | 6 | 8 | 6 | 4
  Week 69 | 0.192 (0.5491) | 0.213 (0.6097) | 0.142 (0.5981) | 0.016 (0.7005) | -0.011 (0.2858)
  Week 87: number analyzed (Participants) | 1 | 6 | 6 | 5 | 2
  Week 87 | 0.517 (0) | 0.164 (0.5377) | 0.247 (0.6591) | 0.086 (0.5132) | -0.044 (0.4264)
  Week 104: number analyzed (Participants) | 1 | 3 | 4 | 4 | 1
  Week 104 | 0.491 (0) | -0.168 (0.4650) | 0.307 (0.3772) | -0.015 (0.5626) | 0.303 (0)

6. Secondary Outcome: Change From Baseline for Mean Daily Glucose Levels Prior to Meals and Bedtime
Description: For each visit, the mean daily glucose levels were calculated over the previous 3-7 days prior to the study visit from blood glucose levels recorded daily prior to meals and bedtime.
Time Frame: Baseline, Weeks 2, 4, 14, 27, 39, 52, 69, 87, and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Alpha1-PI 180 mg/kg/wk, 26 Weeks | 180 mg/kg/wk Alpha1-PI, 13 Weeks | 90 mg/kg/wk Alpha1-PI, 26 Weeks | 90 mg/kg/wk Alpha1-PI, 13 Weeks | Placebo
Number analyzed (Participants) | 15 | 16 | 15 | 15 | 15
mmol/L
  Week 2: number analyzed (Participants) | 11 | 12 | 10 | 11 | 11
  Week 2 | 2.223 (3.6282) | 2.379 (2.7555) | 1.848 (1.1257) | 0.578 (1.6824) | 0.178 (1.5195)
  Week 4: number analyzed (Participants) | 11 | 12 | 10 | 12 | 11
  Week 4 | 2.343 (2.3942) | 1.856 (2.4750) | 2.106 (1.3144) | 0.759 (1.0403) | -0.158 (1.4665)
  Week 14: number analyzed (Participants) | 10 | 9 | 10 | 13 | 12
  Week 14 | 2.812 (2.5953) | 2.200 (2.1283) | 2.852 (3.0376) | 2.337 (3.9732) | -0.053 (1.4368)
  Week 27: number analyzed (Participants) | 7 | 10 | 9 | 9 | 9
  Week 27 | 1.782 (1.7921) | 2.252 (2.8173) | 2.446 (3.2355) | 3.471 (3.1043) | 0.577 (2.1475)
  Week 39: number analyzed (Participants) | 4 | 9 | 8 | 8 | 8
  Week 39 | 1.347 (2.0674) | 3.848 (2.2236) | 4.471 (2.7390) | 3.681 (4.0469) | 1.421 (2.1779)
  Week 52: number analyzed (Participants) | 7 | 11 | 9 | 8 | 8
  Week 52 | 2.995 (1.6703) | 3.067 (2.9160) | 3.242 (3.1636) | 2.723 (4.3749) | 0.616 (2.1868)
  Week 69: number analyzed (Participants) | 5 | 10 | 8 | 6 | 7
  Week 69 | 2.182 (1.3352) | 18.224 (41.1471) | 4.324 (4.4173) | 3.677 (3.7397) | 1.467 (4.2254)
  Week 87: number analyzed (Participants) | 2 | 7 | 7 | 5 | 2
  Week 87 | 3.354 (2.9550) | 3.101 (2.3859) | 3.234 (2.1516) | 3.835 (3.6760) | 4.863 (2.5173)
  Week 104: number analyzed (Participants) | 1 | 4 | 4 | 4 | 3
  Week 104 | 2.545 (0) | 1.867 (2.4532) | 2.390 (1.5429) | 2.283 (6.1064) | 2.431 (1.4519)

ADVERSE EVENTS:
Time Frame: All AEs occurring after subject consent through Week 52 were collected
Description: One subject in the 90 mg/kg/wk Alpha-1 PI, 26 Weeks group prematurely withdrew from the study, did not receive study drug, and was excluded from the safety population.
Arm/Group | Alpha1-PI 180 mg/kg/wk, 26 Weeks | 180 mg/kg/wk Alpha1-PI, 13 Weeks | 90 mg/kg/wk Alpha1-PI, 26 Weeks | 90 mg/kg/wk Alpha1-PI, 13 Weeks | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/16 | 0/14 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 3/16 | 0/14 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 8/16 | 11/14 | 13/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha1-PI 180 mg/kg/wk, 26 Weeks (N=15) | 180 mg/kg/wk Alpha1-PI, 13 Weeks (N=16) | 90 mg/kg/wk Alpha1-PI, 26 Weeks (N=14) | 90 mg/kg/wk Alpha1-PI, 13 Weeks (N=15) | Placebo (N=15)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha1-PI 180 mg/kg/wk, 26 Weeks (N=15) | 180 mg/kg/wk Alpha1-PI, 13 Weeks (N=16) | 90 mg/kg/wk Alpha1-PI, 26 Weeks (N=14) | 90 mg/kg/wk Alpha1-PI, 13 Weeks (N=15) | Placebo (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inner ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 0 (0) | 4 (4) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertrophy (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 3 (5) | 3 (4) | 2 (2)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (9) | 4 (6) | 3 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthroscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 4 (7) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes